CLINICAL TRIAL: NCT01913951
Title: A Phase I Study of Vosaroxin Plus Azacitidine for Patients With Myelodysplastic Syndrome
Brief Title: Vosaroxin and Azacitidine in Treating Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Sunesis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201309091
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — vosaroxin; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (vosaroxin, azacitidine) (Experimental): Patients receive vosaroxin IV over 10 minutes on days 1 and 4 and azacitidine SC or IV over 15 minutes on days 1-7. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vosaroxin; Drug: Azacitidine

INTERVENTIONS:
Drug: vosaroxin — Given IV over 10 minutes on Day 1 and 4
  Other Names: voreloxin
Drug: Azacitidine — Given SC or IV over 15 minutes on days 1-7
  Other Names: Vidaza; Ladakamycin

SUMMARY:
This phase I trial studies the side effects and the best dose of vosaroxin when given together with azacitidine in treating patients with myelodysplastic syndromes. Drugs used in chemotherapy, such as vosaroxin and azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myelodysplastic syndrome and one of the following:

  * Cytopenias requiring red blood cell and/or platelet transfusions or neutropenia (ANC <1 X109/L)
  * IPSS score of INT-1 or higher at screening
  * MDS with excess blasts in transformation as defined by FAB criteria (20-29% bone marrow blasts) or
  * Chronic myelomonocytic leukemia
* Age ≥18 years old
* Adequate renal and hepatic function defined as all of the following:

  * total bilirubin ≤ 2.0 mg/dl, except in cases of Gilbert's disease;
  * AST and ALT ≤2.5 institutional ULN;
  * serum creatinine within normal institutional limits or estimated creatinine clearance ≥60 mL/min/1.73 m2 by the Cockcroft-Gault equation
* ECOG performance status ≤2
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).
* Females must be surgically or biologically sterile or postmenopausal or if of childbearing potential, must agree to use an adequate method of contraception during the study until 30 days after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 30 days after the last treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Patients may have received up to 3 prior cycles of hypomethylator therapy (i.e. decitabine or azacitidine) prior to enrollment and may have received supportive care measures (growth factors, erythropoietin stimulating agents, transfusion, etc.
* Either enrolled in HRPO# 201011766 ("Tissue Acquisition for Analysis of Genetic Progression Factors in Hematologic Diseases"), which facilitates collection of blood, bone marrow, and skin for correlative studies, or consents to collection of blood, bone marrow, and skin as part of this protocol.

Exclusion Criteria:

* Prior treatment with four or more cycles of hypomethylator therapy.
* Receiving concomitant chemotherapy, radiation therapy, or immunotherapy during the duration of treatment on protocol.
* Known seropositivity for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible. Patients who are seropositive for HCV, but have a negative viral load are also eligible. Documentation that the patients have completed a course of therapy for HCV is required and will be obtained.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and/or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-11-22 (Actual); Primary Completion 2016-12-05 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
MTD of vosaroxin in combination with azacitidine | 28 days
  Defined as the highest dose of vosaroxin that results in a DLT in =< 1 of 6 patients graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 4.0

SECONDARY OUTCOMES:
Best response (including hematologic improvement) | At 3 cycles
  According to the modified IWG criteria. Summarized as proportion with 95% confidence intervals.
Best overall response | Up to 7 months
  According to the modified IWG criteria. Summarized as proportion with 95% confidence intervals
Incidence of adverse events | Up to 7 months
  Graded according to NCI CTCAE v. 4.0. summarized by grade, type and patient.
Time to response | Up to 7 months
  According to the modified IWG criteria. Described using Kaplan-Meier models to plot these endpoints and estimate median times with a 95% confidence interval.
Event-free survival | up to 5 years
  From the date of first dose of study drug to date of treatment failure, recurrence, or death due to any cause. Described using Kaplan-Meier models to plot these endpoints and estimate median times with a 95% confidence interval.
Progression-free survival (PFS) | up to 5 years
  From the date of first dose of study drug to disease progression or death from MDS. Described using Kaplan-Meier models to plot these endpoints and estimate median times with a 95% confidence interval.
Disease-free survival (DFS) | up to 5 years
  From the date of first documentation of a complete remission (CR) to date of relapse. Described using Kaplan-Meier models to plot these endpoints and estimate median times with a 95% confidence interval.
Overall survival (OS) | up to 5 years
  Date of first dose of study drug to the date of death from any cause. Described using Kaplan-Meier models to plot these endpoints and estimate median times with a 95% confidence interval.
Biomarkers of response to vosaroxin and azacitidine therapy | Up to 5 years
  Serial estimate of biomarker expression will be plotted and summarized over time using means and standard deviations, possibly on a log scale

CONTACTS AND LOCATIONS:
Overall Officials: Meagan Jacoby, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lancet JE, Ravandi F, Ricklis RM, Cripe LD, Kantarjian HM, Giles FJ, List AF, Chen T, Allen RS, Fox JA, Michelson GC, Karp JE. A phase Ib study of vosaroxin, an anticancer quinolone derivative, in patients with relapsed or refractory acute leukemia. Leukemia. 2011 Dec;25(12):1808-14. doi: 10.1038/leu.2011.157. Epub 2011 Jul 15. PMID 21760592
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu